CLINICAL TRIAL: NCT04532684
Title: Comparison of the Efficacy of Duloxetine and Pregabalin in Patients With Knee Osteoarthritis With Mix Type Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ozgeilleez
Record Dates: First submitted 2020-08-23; First posted 2020-08-31 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2020-05

CONDITIONS: Knee Osteoarthritis
Keywords: Knee osteoartrhritis; Duloxetine; Pregabalin; Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Pain | interventions — Duloxetine Hydrochloride; Pregabalin

STUDY DESIGN:
Intervention Model Description: Randomized prospective clinical trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (Participant, Outcome Assesor)
Oversight: Data Monitoring Committee: No

ARMS (2):
- Duloxetine (Active Comparator): 33 patients received 60 mg/day of duloxetine HCL orally for 12 weeks
  Interventions: Drug: Duloxetine
- Pregabalin (Active Comparator): 33 patients received 300 mg/day of pregabalin orally for 12 weeks
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Duloxetine
  Arms: Duloxetine
Drug: Pregabalin
  Arms: Pregabalin

SUMMARY:
Osteoarthritis (OA) is a common degenerative joint disorder associated with chronic pain at older age.It is known that patients with osteoarthritis experience nociceptive and neuropathic pain to varying degrees. Addition of molecules targeting neuropathic pain to conventional therapy has been shown to improve treatment response in the management of osteoarthritis.The aim of our study is to evaluate the effect of duloxetine and pregabalin on pain, functional capacity, quality of life, depression, anxiety and sleep patterns in knee osteoarthritis.

DETAILED DESCRIPTION:
A total of 66 patients (aged 40-69) with knee osteoarthritis were randomized into two treatment groups to receive either duloxetine 60mg/day or pregabalin 300mg/day. The patients were evaluated before and one month after treatment and three months after treatment using the visual analog scale (VAS-pain), Neuropathic Pain Diagnostic Questionnaire (DN4), Short Form-36 (SF-36) Questionnaire, Western Ontario and McMaster University Osteoarthritis İndeks (WOMAC), Beck Depression Scale (BDS), Beck Anxiety Akalası (BAS), Pittsburg Sleep Quality Index (PSQI).

ELIGIBILITY:
Inclusion Criteria:

* Aged 40-69
* Diagnosed with knee osteoarthritis according to the American College of Rheumatology (ACR) criteria
* Grade 2-3 knee osteoarthritis according to Kellgren-Lawrence grading system
* VAS-pain score: 4 and above
* Neuropathic Pain Diagnostic Questionnaire (DN4) score: 4 and above
* Body mass index value: 40 and below

Exclusion Criteria:

* A history of trauma or surgical operation in the knee region
* Diabetes mellitus
* Fibromyalgia
* Inflammatory rheumatic disease
* Central or peripheral neurological disorder
* Severe cardiac, pulmonary, or malignant disease
* Invasive treatment for knee last 3 months

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Assessing Visual Analog Scale Score Change in Patients | 0.,4., and 12. weeks
  All patients were asked to score the severity of their current knee pain on a 10-cm visual analogue scale (VAS).
Neuropthic Pain Diagnostic Questionnaire (DN4) | 0.,4, and 12. weeks
  There are 10 questions in the DN-4 including 7 questions related to pain quality and 3 questions that investigate the presence of tactile sensation, pinprick sensation, and allodynia. A total score 4/10 indicates neuropathic pain.
Assessing Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Score Change in Patients | 0., 4. and 12. weeks
  The WOMAC consists of 24 questions that assess pain, stiffness, and problems with physical activities. The patient answers all questions on a 5-point Likert-type scale, and the total score ranges from 0 and 96.

SECONDARY OUTCOMES:
Assessing Beck Depression Inventory Score Change in Patients | 0., 4. and 12. weeks
  Symptoms of depression were evaluated by means of the Beck Depression Inventory
Assesing Beck Anxiety Inventory Score Change in Patients | 0.,4.,and 12. weeks
  Current anxiete state of patients was assessed by means of the Beck Anxiety Inventory
Assessing Pittsburgh Sleep Quality Index Score Change in Patients | 0.,4.,and 12. weeks
  Sleep quality assessments were performed by means of the Pittsburgh Sleep Quality Index
Assessing Short Form-36 (SF-36) Questionnaire Score Change in Patients | 0.,4.,and 12. weeks
  The SF-36 has eight subscales and consists of a total of 36 questions. The subscales are vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health. A score of 0 is equivalent to maximum disability (poor quality of life), and a score of 100 is equivalent to no disability (good quality of life).

CONTACTS AND LOCATIONS:
Overall Officials: Özge Gülsüm İlleez, M.D, Principal Investigator — Fatih Sultan Mehmet Training and Research Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leaney AA, Lyttle JR, Segan J, Urquhart DM, Cicuttini FM, Chou L, Wluka AE. Antidepressants for hip and knee osteoarthritis. Cochrane Database Syst Rev. 2022 Oct 21;10(10):CD012157. doi: 10.1002/14651858.CD012157.pub2. PMID 36269595